CLINICAL TRIAL: NCT06204601
Title: The Effect Of Education Given According to Meleıs' Transitional Theory on The Level of Self-Effectiveness With Anxiety and Depression to Patients With Pacemaker: A Single-Blind Randomized Controlled Study
Brief Title: The Effect Of Education Given According to Meleıs' Transitional Theory to Patients With Pacemaker
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hacer Gok Ugur, Associate Professor., Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2Ordu
Record Dates: First submitted 2023-11-01; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Educational Activities
Keywords: Pacemaker,; Meleis Transition Theory,; Education,; Self-Efficacy,; Anxiety, Depression,; Nursing
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: Trial model with pretest posttest control group
Who Masked: Participant
Masking Description: Block randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental group
  Interventions: Other: Education According to Meleis' Transitional Theory to Patients With Pacemaker
- Control group (No Intervention): Control group

INTERVENTIONS:
Other: Education According to Meleis' Transitional Theory to Patients With Pacemaker — Patients in the experimental group will be trained according to Meleis's Transition Theory.
  Arms: Experimental group

SUMMARY:
This study will be carried out to determine the effect of training given according to Meleis's Transition Theory to patients with pacemaker implantation on anxiety, depression and self-efficacy levels.

DETAILED DESCRIPTION:
This study will be carried out to determine the effect of training given according to Meleis's Transition Theory to patients with pacemaker implantation on anxiety, depression and self-efficacy levels.

Hypotheses of the Research H01: Training given to patients with pacemaker implantation according to Meleis's Transition Theory does not affect the anxiety and depression levels of the patients.

H11: Training given according to Meleis's Transition Theory to patients with pacemaker implants reduces the anxiety and depression levels of patients.

H02: Training given to patients with pacemaker implantation according to Meleis's Transition Theory does not affect the self-efficacy level of the patients.

H12: Training given to patients with pacemakers according to Meleis's Transition Theory increases the self-efficacy level of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pacemaker implantation,
* Ages 18 and over,
* The one who is literate,
* Open to communication and collaboration,
* Patients who volunteer to participate in the study will be included in the study.

Exclusion Criteria:

* Not oriented to person, place and time,
* Hearing loss,
* Cannot understand and speak Turkish and
* Patients who do not want to continue the study will be excluded from the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | month 1
  The scale was developed by Zigmond and Snaith (1983) to determine the risk of anxiety and depression in patients and was translated into Turkish by Aydemir et al. Adapted from (1997). It consists of a total of 14 questions, odd numbered questions measure anxiety, and even numbered questions measure depression. The scale provides four-point Likert type measurement. In scoring; Items 1, 3, 5, 6, 8, 10, 11 and 13 are in the format 3,2,1,0, 2, 4, 7, 9, 12 and 14. The items are scored as 0,1,2,3. By summing the 1st, 3rd, 5th, 7th, 9th, 11th and 13th items of the anxiety subscale of the scale, the depression subscale; It is calculated by adding the 2nd, 4th, 6th, 8th, 10th, 12th and 14th items. The cut-off score for the anxiety subscale is 10/11 and for the depression subscale is 7/8. Accordingly, areas above these scores are considered at risk.

SECONDARY OUTCOMES:
Self-Efficacy Scale in Chronic Diseases | month 1
  The scale was developed by Lorig et al. (1996) in 1996 to measure the self-efficacy perceptions of individuals with chronic diseases and was adapted into Turkish by Ceyhan and Ünsal (2017). The scale generally consists of three main concepts and a total of 10 sub-dimensions. In order to realize the first concept, "Self-management behaviors", under the heading of PE; The sub-dimensions include doing regular sports, getting information about the disease, getting help from society, family and friends, and communicating with the doctor. The scale is answered in Likert type, increasing from 0 to 10, which determines the perception of PE. The number 0 on the scale represe

CONTACTS AND LOCATIONS:
Overall Officials: Hacer GÖK UĞUR, Asos.Prof., Principal Investigator — Ordu Univercity
Locations (2):
- Turkey (Türkiye) (2):
  - Hacer GOK UGUR, Ordu, Altınordu
  - Hacer GÖK UĞUR, Ordu

IPD SHARING:
Plan to Share IPD: No